CLINICAL TRIAL: NCT00427622
Title: A Trial to Examine the Accuracy of an Ambulatory Sternal Skin Conductance Recording Tool to Measure Hot Flashes
Brief Title: Skin Conduction Device for Measuring Hot Flashes in Postmenopausal Women With Hot Flashes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Diagnostic
Other Study IDs: MC05CC; MC05CC (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2007-06

CONDITIONS: Hot Flashes
Keywords: hot flashes
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: physiologic testing

SUMMARY:
RATIONALE: Measuring how often hot flashes occur in postmenopausal women may be done by using a skin conduction device or by using a diary.

PURPOSE: This clinical trial is comparing a skin conduction device with a hot flash diary as a way of measuring hot flashes in postmenopausal women with hot flashes.

DETAILED DESCRIPTION:
OBJECTIVES:

* Correlate hot flash frequency, as measured by an ambulatory sternal skin conductance measuring and recording tool, with patient-recorded hot flash frequency using a hot flash diary in postmenopausal women with hot flashes.
* Determine the comfort, obtrusiveness, and feasibility of using the skin conductance recording tool for measuring hot flashes when worn daily for five weeks in these patients.

OUTLINE: Patients wear an ambulatory sternal skin conductance hot flash device continuously for 5 weeks.

Patients complete hot flash diaries once daily for 5 weeks. Patients also complete the Comfort, Bother, and Weight Questionnaire at the end of week 5.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of bothersome hot flashes, defined by their occurrence of ≥ 4 times/day

  * Daily hot flashes have been present for ≥ 1 month

PATIENT CHARACTERISTICS:

* Female
* Postmenopausal
* ECOG performance status 0-1
* No history of allergic or other adverse reactions to adhesives
* No other medical condition known to cause sweating and/or flushing
* Willing to record hot flashes in a hot flash diary daily for 5 weeks
* Willing to wear a skin conductance device 24 hours a day for 5 weeks
* No implanted pacemakers or metal implants
* No reliance on other electronic devices for regular monitoring (i.e., insulin pumps or blood pressure monitors)

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2006-05; Primary Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Correlation of hot flash frequency, as measured by an ambulatory sternal skin conductance measuring and recording tool, with patient-recorded hot flash frequency using a hot flash diary
Comfort, obtrusiveness, and feasibility of using the skin conductance recording tool

CONTACTS AND LOCATIONS:
Overall Officials: Debra Barton, RN, PhD, AOCN, FAAN, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States